CLINICAL TRIAL: NCT07130279
Title: The Effect of Post-Isometric Relaxation Technique on Cervical Range of Motion, Mandibular Mobility, Head Anterior Tilt, and Kyphotic Posture in Individuals With Temporomandibular Joint Dysfunction
Brief Title: Post-Isometric Relaxation in Temporomandibular Disorders
Acronym: PIR-TMD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sanem ŞENER (Other)
Responsible Party: Sponsor-Investigator, Sanem ŞENER, Assistant Professor, Bulent Ecevit University
Organization: Bulent Ecevit University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TME-PIR-2024-01
Record Dates: First submitted 2025-08-11; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Temporomandibular Joint Disorders; Myofascial Pain Syndromes; Mandibular Dysfunction
Keywords: Temporomandibular Joint Dysfunction; Post-Isometric Relaxation; range of motion
MeSH Terms: conditions — Temporomandibular Joint Disorders; Myofascial Pain Syndromes | interventions — Methods

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned into two parallel groups: the experimental group will receive postural exercises combined with the Post-Isometric Relaxation (PIR) technique, while the control group will receive postural exercises only. Both groups will follow the intervention protocol three times per week for six weeks, with no crossover between groups.
Who Masked: Outcomes Assessor
Masking Description: This is a single-masked trial in which the outcomes assessor is blinded to group allocation. The assessor responsible for measuring cervical range of motion, mandibular mobility, head anterior tilt, and thoracic kyphosis index will not be informed of the participants' assigned intervention group
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Arm: Postural Exercises + Post-Isometric Relaxation (PIR) Technique (Experimental): Participants in this group will perform a standardized postural exercise program targeting cervical and thoracic regions, three times per week for six weeks. In addition, the Post-Isometric Relaxation (PIR) technique will be applied to the jaw muscles during each session, following a standardized manual therapy protocol to reduce muscle tension and improve mandibular mobility.
  Interventions: Behavioral: Postural Exercises + Post-Isometric Relaxation (PIR) Technique; Behavioral: Postural Exercises
- Control Arm: Postural Exercises Only (Active Comparator): Participants in this group will perform the same standardized postural exercise program targeting cervical and thoracic regions, three times per week for six weeks, without the addition of the PIR technique.
  Interventions: Behavioral: Postural Exercises

INTERVENTIONS:
Behavioral: Postural Exercises + Post-Isometric Relaxation (PIR) Technique — Participants will perform a standardized postural exercise program (strengthening, stretching, and mobility exercises for the cervical and thoracic regions) three times per week for six weeks. In addition, the Post-Isometric Relaxation (PIR) technique will be applied to jaw muscles during each session to reduce muscle tension and improve mandibular mobility.
  Arms: Experimental Arm: Postural Exercises + Post-Isometric Relaxation (PIR) Technique
Behavioral: Postural Exercises — Participants will perform a standardized postural exercise program designed to improve cervical and thoracic mobility and postural alignment. The program will include strengthening, stretching, and mobility exercises targeting the cervical spine, thoracic spine, and related musculature. Each session will last approximately 30-40 minutes and will be conducted three times per week for six weeks under the supervision of a trained therapist.

SUMMARY:
This planned randomized, single-blind clinical trial will investigate the effects of adding the Post-Isometric Relaxation (PIR) technique to a standard postural exercise program in individuals with moderate to severe temporomandibular joint dysfunction (TMD). Forty volunteers aged 18-25 years will be recruited and randomly assigned to either an experimental group (postural exercises + PIR) or a control group (postural exercises only). The intervention will be delivered three times per week for six weeks. Primary outcomes will include cervical range of motion, mandibular mobility, head anterior tilt, and thoracic kyphosis index, measured before and after the intervention. The study aims to determine whether PIR provides additional benefits to standard postural exercises in improving jaw and neck function and postural alignment in young adults with TMD.

DETAILED DESCRIPTION:
Temporomandibular joint dysfunction (TMD) is a common musculoskeletal condition characterized by jaw pain, limited mouth opening, and joint sounds, often accompanied by postural deviations such as forward head posture and thoracic kyphosis. Conservative treatments, including postural exercises and manual therapy, are recommended to improve jaw and neck function and reduce symptoms.

The Post-Isometric Relaxation (PIR) technique is a manual therapy method that uses gentle isometric contractions followed by passive stretching to reduce muscle tension and increase mobility. While PIR has been shown to improve masticatory muscle function, its combined use with postural exercises in TMD management has not been fully evaluated.

In this planned study, forty volunteers aged 18-25 years with moderate or severe TMD (diagnosed using the Fonseca Anamnestic Questionnaire) will be recruited. Participants will be randomly assigned into two groups:

Experimental group: Postural exercise program + PIR technique

Control group: Postural exercise program only

The postural exercise program will include strengthening, stretching, and mobility exercises for the cervical and thoracic regions, performed three times per week for six weeks. In the experimental group, the PIR technique will be applied to jaw muscles according to a standardized protocol.

Outcome measures will include:

Cervical range of motion (flexion, extension, lateral flexion, rotation) measured with a goniometer

Mandibular mobility (depression, lateral deviation, protrusion) measured with a caliper

Head anterior tilt (chin-sternum distance, occiput-wall distance)

Thoracic kyphosis index measured with a flexicurve

Assessments will be conducted before the intervention and after the six-week program. The primary hypothesis is that the addition of PIR to postural exercises will produce greater improvements in cervical and mandibular mobility than postural exercises alone.

This trial is expected to provide new evidence for combining manual therapy with exercise in the management of TMD in young adults and may help guide future rehabilitation strategies.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 25 years
* Diagnosis of moderate or severe temporomandibular joint dysfunction (TMD) according to the Fonseca Anamnestic Questionnaire
* Presence of TMD symptoms for at least 6 months
* No TMD treatment received within the last 6 months
* Presence of chewing muscle pain for at least 6 months
* Able and willing to participate in the study and follow the exercise program
* Signed informed consent form

Exclusion Criteria:

* History of jaw or facial trauma within the past year
* History of temporomandibular joint surgery
* Presence of systemic rheumatologic, neurological, or musculoskeletal disorders affecting the jaw, neck, or spine
* Pregnancy
* Current participation in another clinical trial
* Inability to perform the exercise program due to medical or physical limitations
* Refusal to provide informed consent

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-08-11 (Estimated); Primary Completion 2025-09-22 (Estimated); Study Completion 2025-09-25 (Estimated)

PRIMARY OUTCOMES:
Change in mandibular depression (mouth opening) | Baseline and after 6 weeks of intervention
  The distance between the upper and lower central incisors during maximal mouth opening will be measured in millimeters using a caliper.
Change in cervical range of motion | Baseline and after 6 weeks of intervention
  Cervical range of motion will be measured in degrees using a goniometer. Movements assessed will include flexion, extension, right and left lateral flexion, and right and left rotation.
Change in mandibular lateral deviation (right and left) | Baseline and after 6 weeks of intervention
  The horizontal movement of the lower jaw to the right and left will be measured in millimeters using a caliper.
Change in mandibular protrusion | Baseline and after 6 weeks of intervention
  The anterior translation of the mandible will be measured in millimeters using a caliper.
  Outcome Measure: Change in head anterior tilt - chin-sternum distance
Change in head anterior tilt - chin-sternum distance | Baseline and after 6 weeks of intervention
  The vertical distance from the midpoint of the chin to the superior border of the sternum will be measured in centimeters with a measuring tape.
Change in head anterior tilt - occiput-wall distance | Baseline and after 6 weeks of intervention
  The distance between the occiput and the wall will be measured in centimeters while the participant stands in a natural posture against the wall.
Change in thoracic kyphosis index | Baseline and after 6 weeks of intervention
  Thoracic kyphosis will be evaluated using a flexicurve ruler to measure curvature from C7 to T12. The thoracic kyphosis index will be calculated as (thoracic width / thoracic length) × 100.

CONTACTS AND LOCATIONS:
Overall Officials: Sanem ŞENER, Principal Investigator — Zonguldak Bulent Ecevit University

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared because the study's ethics committee approval does not include provisions for external sharing of raw participant-level data. Data will be stored securely at Yeniyüzyıl University and will only be accessible to the research team for purposes of analysis and reporting